CLINICAL TRIAL: NCT02028884
Title: A Multicenter, Randomized, Addition to Baseline Treatment, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Satralizumab (SA237) in Patients With Neuromyelitis Optica (NMO) and NMO Spectrum Disorder (NMOSD)
Brief Title: Efficacy and Safety Study of Satralizumab (SA237) as Add-on Therapy to Treat Participants With Neuromyelitis Optica (NMO) and NMO Spectrum Disorder (NMOSD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN40898; 2013-003752-21 (EudraCT Number); SA-307JG (Other: Chugai Pharmaceutical)
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Neuromyelitis Optica (NMO); NMO Spectrum Disorder (NMOSD)
MeSH Terms: conditions — Neuromyelitis Optica | interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Satralizumab + Baseline Treatment (Experimental): Participants randomized to this arm for the double-blind period will receive satralizumab in addition to baseline treatment. The double-blind period ends when either the participant has a treated relapse or the total number of protocol-defined relapses confirmed by the Clinical Endpoint Committee (CEC) reaches 26. In the open-label extension period, the participant will receive (with or without baseline treatment) an SC injection of satralizumab at Weeks 0, 2, and 4, and Q4W thereafter, with the last study drug administration on or before 31 December 2021.
  Interventions: Drug: Satralizumab; Drug: Baseline Treatment
- Placebo + Baseline Treatment (Placebo Comparator): Participants randomized to this arm for the double-blind period will receive placebo in addition to baseline treatment.The double-blind period ends when either the participant has a treated relapse or the total number of protocol-defined relapses confirmed by the Clinical Endpoint Committee (CEC) reaches 26. In the open-label extension period, the participant will receive (with or without baseline treatment) an SC injection of satralizumab at Weeks 0, 2, and 4, and Q4W thereafter, with the last study drug administration on or before 31 December 2021.
  Interventions: Drug: Placebo; Drug: Baseline Treatment

INTERVENTIONS:
Drug: Satralizumab — Satralizumab will be administered subcutaneously (SC) at Weeks 0, 2, and 4, and thereafter once every 4 weeks (Q4W).
  Other Names: SA237; RG6168; RO5333787
  Arms: Satralizumab + Baseline Treatment
Drug: Placebo — Placebo will be administered subcutaneously (SC) at Weeks 0, 2, and 4, and thereafter once every 4 weeks (Q4W).
  Arms: Placebo + Baseline Treatment
Drug: Baseline Treatment — As specified in the protocol, one of the following drugs at a stable dose is required as monotherapy for baseline treatment during the double-blind period: azathioprine (AZA); mycophenolate mofetil (MMF); or oral corticosteroids (CS). For participants aged 12 to 17 years at the time of informed consent, baseline treatment with AZA or MMF in combination with oral CS is also permitted. Change or termination of baseline treatment is only permitted during the open-label extension period.

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, pharmacodynamic, pharmacokinetic, and immunogenic profiles of satralizumab, compared with placebo, in addition to baseline immunosuppressive treatment in participants with NMO and NMOSD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed as having either neuromyelitis optica (NMO) or NMO spectrum disorder (NMOSD), defined as the following:

   1. NMO as defined by Wingerchuk et al. 2006 criteria (requires all of the following 3 criteria: I. Optic neuritis, II. Acute myelitis, III. At least two of three supportive criteria: Contiguous spinal cord lesion identified on a magnetic resonance imaging (MRI) scan extending over 3 vertebral segments; Brain MRI not meeting diagnostic criteria for multiple sclerosis (MS); NMO-IgG seropositive status)
   2. NMOSD as defined by either of the following Wingerchuk 2007 criteria with anti-AQP4 antibody (Ab) seropositive status at screening (i. Idiopathic single or recurrent events of longitudinally extensive myelitis [≥3 vertebral segment spinal cord MRI lesion]; ii. Optic neuritis: recurrent or simultaneous bilateral); For patients aged 12 to 17 years, a minimum of 4 patients should be positive for anti-AQP4Ab status at screening
2. Clinical evidence of at least 2 documented relapses (including first attack) in the last 2 years prior to screening, at least one of which has occurred in the 12 months prior to screening
3. EDSS score from 0 to 6.5 inclusive at screening
4. Age 12 to 74 years, inclusive at the time of informed consent
5. One of the following baseline treatments must be at stable dose as a monotherapy for 8 weeks prior to baseline: Azathioprine; Mycophenolate mofetil; Oral corticosteroids. For participants aged 12 to 17 years, either of the following baseline treatments for relapse prevention can be allowed: Azathioprine + oral corticosteroids; Mycophenolate mofetil + oral corticosteroids
6. Ability and willingness to provide written informed consent and to comply with the requirements of the protocol

For adolescents who may be enrolled after the end of the double-blind period, the inclusion criterion 2 is as follows (other criteria are same): Clinical evidence of at least 2 documented relapses (including first attack) prior to screening.

Exclusion Criteria:

Exclusion criteria related to previous or concomitant therapy:

1. Any previous treatment with IL-6 inhibitory therapy (e.g. tocilizumab), alemtuzumab, total body irradiation or bone marrow transplantation at any time
2. Any previous treatment with anti-CD20, eculizumab, belimumab, interferon, natalizumab, glatiramer acetate, fingolimod, teriflunomide or dimethyl fumarate within 6 months prior to baseline
3. Any previous treatment with anti-CD4, cladribine or mitoxantrone within 2 years prior to baseline
4. Treatment with any investigational agent within 3 months prior to baseline

   Exclusions for general safety:
5. Pregnancy or lactation
6. For patients of reproductive potential, a positive result from a serum pregnancy test at screening, or not willing to use reliable means of contraception (physical barrier [patient or partner] in conjunction with a spermicidal product, contraceptive pill, patch, injectables, intrauterine device or intrauterine system) during the treatment period and for at least 3 months after the last dose of study drug
7. Any surgical procedure (except for minor surgeries) within 4 weeks prior to baseline
8. Evidence of other demyelinating disease or progressive multifocal leukoencephalopathy (PML)
9. Evidence of serious uncontrolled concomitant diseases that may preclude patient participation, such as: other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency
10. Known active infection (excluding fungal infections of nail beds or caries dentium) within 4 weeks prior to baseline
11. Evidence of chronic active hepatitis B or C
12. History of drug or alcohol abuse within 1 year prior to baseline
13. History of diverticulitis that, in the Investigator's opinion, may lead to increased risk of complications such as lower gastrointestinal perforation
14. Evidence of active tuberculosis (TB; excluding patients receiving chemoprophylaxis for latent TB infection)
15. Evidence of active interstitial lung disease
16. Receipt of any live or live attenuated vaccine within 6 weeks prior to baseline
17. History of malignancy within the last 5 years, including solid tumors, hematologic malignancies and in situ carcinoma (except basal cell and squamous cell carcinomas of the skin, or in situ carcinoma of the cervix uteri that have been completely excised and cured)
18. History of severe allergic reaction to a biologic agent (e.g. shock, anaphylactic reactions)
19. Active suicidal ideation within 6 months prior to screening, or history of suicide attempt within 3 years prior to screening
20. Following laboratory abnormalities at screening*.

    1. White blood cells (WBC) <3.0 x10^3/microliter (μL)
    2. Absolute neutrophil count (ANC) <2.0 x10^3/μL
    3. Absolute lymphocyte count <0.5 x10^3/μL
    4. Platelet count <10 x 10^4/μL
    5. Aspartate aminotransferase (AST) or alanine aminotranferase (ALT) >1.5 times the upper limit of normal (ULN) * If retest is conducted, the last value of retest before randomization must meet study criteria.

For adolescents who may be enrolled after the end of the double-blind period, the annotation in the exclusion criterion 20 is as follows (other criteria are same): * If retest is conducted, the last value of retest before baseline must meet study criteria

Ages: 12 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- Children's Hospital of Alabama, Birmingham, Alabama, United States
- Hopital de Hautepierre CHRU de Strasbourg, Strasbourg, France
- Germany (3):
  - NeuroCure Clinical Research Center (NCRC), Berlin
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Heinrich-Heine Universitätsklinik Düsseldorf, Düsseldorf
- Jahn Ferenc Dél-Pesti Kórház, Budapest, Hungary
- Italy (4):
  - Azienda Ospedaliera Sant'Andrea-Universitr di Roma La Sapien, Rome, Lazio
  - Ospedale San Raffaele, Milan, Lombardy
  - PO G.Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania, Sicily
  - Fond. Ist. S. Raffaele - giglio, Cefalù, Sicily
- Japan (10):
  - Juntendo University Hospital; Neurology, Bunkyō City
  - Kyushu University Hospital; Neurology, Fukuoka
  - Fukushima Medical University Hospital; Neurology, Fukushima
  - Kagoshima University Medical And Dental Hospital; Neurology and Geriatorics, Kagoshima
  - Niigata University Medical and Dental Hospital; Neurology, Niigata
  - Kindai University Hospital; Neurology, Osaka
  - Tohoku University Hospital; Neurology, Sendai
  - Tokyo Women's Medical University Hospital; Neurology, Shinjuku-ku
  - Osaka University Hospital; Neurology, Suita
  - National Center of Neurology and Psychiatry, Tokyo
- Poland (7):
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice
  - M.A. - LEK A. M. Maciejowscy SC. Centrum Terapii SM, Katowice
  - Centrum Medyczne Dendryt, Katowice
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Szpital Kliniczny im. H.Swiecickiego UM w Poznaniu, Późna
  - Samodzielny Publiczny Centralny Szpital Klinicznyi, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico San Carlos; Servicio de Nefrologia, Madrid
- Taiwan (5):
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Neurology, Kwei Shen
  - China Medical University Hospital; Neurology - Taichung, Taichung
  - National Cheng Kung University Hospital; Neurology, Tainan
  - National Taiwan University Hospital; Neurology, Taipei
  - Taipei Veterans General Hospital-Neurology, Taipei
- Ukraine (2):
  - Kharkivska miska dytiacha likarnia # 5, Kharkiv, Kharkiv Governorate
  - KZ "Dnipropetrovska oblasna dytiacha klinichna likarnia" DOR, Dnipropetrovsk, Tavria Okruha
- United Kingdom (4):
  - University Hospital of Wales; Dept of Neurology, Cardiff
  - John Radcliffe Hospital; Neurosciences, Chinnor
  - The National Hospital for Neurology & Neurosurgery, London
  - Great Ormond Street Hospital For Children; Neurology, London

REFERENCES:
- [Derived] Bennett JL, Fujihara K, Saiz A, Traboulsee AL, Greenberg BM, Weinshenker BG, Patti F, Kleiter I, Palace J, De Seze J, Evans R, Blondeau K, Klingelschmitt G, Vodopivec I, Rahim M, Yamamura T. Long-Term Efficacy and Safety of Satralizumab in Patients With Neuromyelitis Optica Spectrum Disorder From the SAkuraMoon Open-Label Extension Study. Neurol Neuroimmunol Neuroinflamm. 2025 Sep;12(5):e200450. doi: 10.1212/NXI.0000000000200450. Epub 2025 Jul 31. PMID 40743487
- [Derived] Greenberg BM, Fujihara K, Weinshenker B, Patti F, Kleiter I, Bennett JL, Palace J, Blondeau K, Burdeska A, Ngwa I, Klingelschmitt G, Triyatni M, Yamamura T. Analysis of infection rates in neuromyelitis optica spectrum disorder: Comparing satralizumab treatment in SAkuraMoon, post-marketing, and US-based health claims data. Mult Scler Relat Disord. 2025 Jul;99:106444. doi: 10.1016/j.msard.2025.106444. Epub 2025 Apr 19. PMID 40288333
- [Derived] Kleiter I, Traboulsee A, Palace J, Yamamura T, Fujihara K, Saiz A, Javed A, Mayes D, Budingen HV, Klingelschmitt G, Stokmaier D, Bennett JL. Long-term Efficacy of Satralizumab in AQP4-IgG-Seropositive Neuromyelitis Optica Spectrum Disorder From SAkuraSky and SAkuraStar. Neurol Neuroimmunol Neuroinflamm. 2022 Dec 8;10(1):e200071. doi: 10.1212/NXI.0000000000200071. Print 2023 Jan. PMID 36724181
- [Derived] Yamamura T, Weinshenker B, Yeaman MR, De Seze J, Patti F, Lobo P, von Budingen HC, Kou X, Weber K, Greenberg B. Long-term safety of satralizumab in neuromyelitis optica spectrum disorder (NMOSD) from SAkuraSky and SAkuraStar. Mult Scler Relat Disord. 2022 Oct;66:104025. doi: 10.1016/j.msard.2022.104025. Epub 2022 Jul 5. PMID 36007339
- [Derived] Yamamura T, Kleiter I, Fujihara K, Palace J, Greenberg B, Zakrzewska-Pniewska B, Patti F, Tsai CP, Saiz A, Yamazaki H, Kawata Y, Wright P, De Seze J. Trial of Satralizumab in Neuromyelitis Optica Spectrum Disorder. N Engl J Med. 2019 Nov 28;381(22):2114-2124. doi: 10.1056/NEJMoa1901747. PMID 31774956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the double-blind (DB) period up to the primary clinical cut-off date (06 June 2018) and in the Open-label Extension Period until the final clinical cut-off date (23-Dec-2021). All ongoing patients have been offered to transition to the WN42349 study
Groups:
- Placebo + Baseline Treatment, Then Satralizumab: Participants received matching placebo, subcutaneous (SC) at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period up to protocol-defined relapse or treated relapse in addition to baseline treatment. Following the DB period all participants received satralizumab 120 mg SC injection (with or without baseline treatment) at Weeks 0, 2 and 4, and Q4W thereafter up to the clinical cut-off date (CCOD). At the CCOD, participants who had not experienced a relapse during the DB period were invited to initiate satralizumab 120 mg SC injection (with or without baseline treatment at Weeks 0, 2 and 4, and Q4W thereafter) after 4 weeks from their last study treatment dose in the DB period.
- Satralizumab + Baseline Treatment, Then Satralizumab: Participants received satralizumab 120 mg SC injection at Weeks 0, 2 and 4, and Q4W thereafter throughout the DB period up to protocol-defined relapse or treated relapse in addition to baseline treatment. Following the DB period all participants received satralizumab 120 mg SC injection (with or without baseline treatment) at Weeks 0, 2 and 4, and Q4W thereafter up to the CCOD. At the CCOD, participants who had not experienced a relapse during the DB period were invited to continue satralizumab 120 mg SC injection (with or without baseline treatment at Weeks 0, 2 and 4, and Q4W thereafter) after 4 weeks from their last study treatment dose in the DB period.
- SA237 - Enrolled in Open-Label: In the open-label extension period, the participant received an SC injection of satralizumab at Weeks 0,2, and 4, and Q4W thereafter, in addition to baseline treatment
Period: Double-blind Period
Arm/Group | Placebo + Baseline Treatment, Then Satralizumab | Satralizumab + Baseline Treatment, Then Satralizumab | SA237 - Enrolled in Open-Label
Started | 42 | 42 | 0
Completed (Double-blind period) | 32 | 39 | 0
Not Completed | 10 | 3 | 0
Not completed — Adverse Event | 5 | 3 | 0
Not completed — Eligibility Violation | 1 | 0 | 0
Not completed — Non-Compliance With Study Drug | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: Open-label Extension Period
Arm/Group | Placebo + Baseline Treatment, Then Satralizumab | Satralizumab + Baseline Treatment, Then Satralizumab | SA237 - Enrolled in Open-Label
Started | 32 | 39 | 1
Completed (Open-label extension period) | 23 | 31 | 1
Not Completed | 9 | 8 | 0
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Refused Treatment/Did Not Cooperate | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 0
Not completed — Switched to another treatment option | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized to the treatment groups.
Groups:
- Placebo + Baseline Treatment: Participants received matching placebo, subcutaneous (SC) at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period up to protocol-defined relapse or treated relapse in addition to baseline treatment. Following the DB period all participants received satralizumab 120 mg SC injection (with or without baseline treatment) at Weeks 0, 2 and 4, and Q4W thereafter up to the clinical cut-off date (CCOD). At the CCOD, participants who had not experienced a relapse during the DB period were invited to initiate satralizumab 120 mg SC injection (with or without baseline treatment at Weeks 0, 2 and 4, and Q4W thereafter) after 4 weeks from their last study treatment dose in the DB period.
- Satralizumab + Baseline Treatment: Participants received satralizumab 120 mg SC injection at Weeks 0, 2 and 4, and Q4W thereafter throughout the DB period up to protocol-defined relapse or treated relapse in addition to baseline treatment. Following the DB period all participants received satralizumab 120 mg SC injection (with or without baseline treatment) at Weeks 0, 2 and 4, and Q4W thereafter up to the CCOD. At the CCOD, participants who had not experienced a relapse during the DB period were invited to continue satralizumab 120 mg SC injection (with or without baseline treatment at Weeks 0, 2 and 4, and Q4W thereafter) after 4 weeks from their last study treatment dose in the DB period.
- Total: Total of all reporting groups
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment | SA237 - Enrolled in Open-Label | Total
Number analyzed (Participants) | 42 | 42 | 1 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (12.00) | 40.2 (16.3) | 16 (NA) — Only one participant in the arm | 41.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 1 | 79
  Male | 2 | 4 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 40 | 42 | 1 | 83
  Not Stated | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18 | 18 | 0 | 36
  Black or African American | 2 | 0 | 0 | 2
  White | 21 | 24 | 0 | 45
  Other | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to First Protocol-Defined Relapse (TFR) in the Double-Blind Period
Description: TFR was defined as time from randomization to first occurrence of relapse in the DB period. Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neurological neuromyelitis optica (NMO) or neuromyelitis optica spectrum disorder (NMOSD) as adjudicated by an independent clinical endpoint committee (CEC). Symptoms had to persist for >24 hours and not be attributable to confounding clinical factors (e.g., fever, infection, injury, change in mood, adverse reactions to medications). New or worsening neurological symptoms that occurred < 31 days following onset of a protocol-defined relapse were considered part of same relapse (i.e., if 2 relapses had onset days that were 30 days of one another, they were counted only as 1 relapse), and onset date used in analysis was the date of first relapse.
Time Frame: Up to Week 224
Population: ITT population included all participants randomized to the treatment groups. For participants who had not relapsed, the TFR was censored on the date of end of the DB period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
weeks | 120.6 [37.0 to NA] — Upper limit of confidence interval (CI) was not reached due to low number of participants with events. | NA [NA to NA] — Median was not reached due to low number of participants with events. Lower and upper limit of CI was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Placebo + Baseline Treatment vs Satralizumab + Baseline Treatment; Stratified by Baseline annualized relapse rate (ARR: 1, > 1) and geographic region (Asia, EU/Other); Test type: Superiority; p = 0.0184, Log Rank; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.16 to 0.88]

2. Secondary Outcome: Change From Baseline at Week 24 in the Visual Analogue Scale (VAS) Score for Pain During the DB Period
Description: The VAS is a subjective measure of pain consisting of a 100 mm line with two endpoints representing 0 = "no pain" and 100 = "pain as bad as it could be". Participants rated their pain by placing a mark on the line corresponding to their current level of pain. The distance along the line from the "no pain" marker was measured with a ruler giving a pain score out of 100. A higher score indicated more pain and lower scores reflected a better health state. A negative change from baseline indicates an improvement. ANCOVA was used for analysis to report the adjusted mean and standard error (SE).
Time Frame: Baseline, Week 24
Population: ITT population included all participants randomized to the treatment groups. Number analyzed is the number of participants with data available for analyses at the given timepoint. Missing data were imputed by baseline observation carried forward (BOCF) method.
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 34.619 (4.026) | 27.561 (4.399)
  Change from Baseline at Week 24 | -3.505 (2.357) | 2.871 (2.391)
Statistical Analysis 1: Comparison: Placebo + Baseline Treatment vs Satralizumab + Baseline Treatment; Test type: Superiority; p = 0.0602, ANCOVA; ANCOVA model: treatment group as fixed effect and baseline measurements, prior therapy, most recent attack (first attack/relapse) as covariates; Mean Difference (Final Values) = 6.376, 95% CI 2-sided [-0.280 to 13.033], Standard Error of Mean 3.344

3. Secondary Outcome: Change From Baseline at Week 24 in the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Score During the DB Period
Description: The FACIT Fatigue scale is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days. As each of the 13 items of the scale ranges from 0-4, the range of possible scores was computed using FACIT scoring algorithm as 0-52, where 0 is the worst possible score and 52 the best which indicated less fatigue. A positive change from baseline indicates an improvement. ANCOVA was used for analysis to report the adjusted mean and SE.
Time Frame: Baseline, Week 24
Population: ITT population included all participants randomized to the treatment groups. Number analyzed is the number of participants with data available for analyses at the given timepoint. Missing data was imputed using BOCF method
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 33.857 (1.746) | 34.732 (1.646)
  Change from Baseline at Week 24 | 2.234 (0.943) | 0.145 (0.963)
Statistical Analysis 1: Comparison: Placebo + Baseline Treatment vs Satralizumab + Baseline Treatment; Test type: Superiority; p = 0.1224, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.089, 95% CI 2-sided [-4.752 to 0.574], Standard Error of Mean 1.338

4. Secondary Outcome: Relapse-Free Rate During the DB Period
Description: Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neurological neuromyelitis optica (NMO) or neuromyelitis optica spectrum disorder (NMOSD). Symptoms had to persist for >24 hours and not be attributable to confounding clinical factors (e.g., fever, infection, injury, change in mood, adverse reactions to medications). New or worsening neurological symptoms that occurred < 31 days following onset of a protocol-defined relapse were considered part of same relapse (i.e., if 2 relapses had onsets within 30 days of one another, they were counted as 1), and onset date used in analysis was the date of first relapse.
Time Frame: Up to Week 216
Population: ITT population included all participants randomized to the treatment groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 34 | 37
percentage of participants
  Week 12 | 89.86 | 94.99
  Week 24 | 84.41 | 88.86
  Week 36 | 69.49 | 88.86
  Week 48 | 66.02 | 88.86
  Week 72 | 58.68 | 81.46
  Week 96 | 58.68 | 77.58
  Week 120 | 54.17 | 73.70
  Week 144 | 49.24 | 73.70
  Week 168 | 43.77 | 73.70
  Week 192: number analyzed (Participants) | 0 | 37
  Week 192 |  | 73.70
  Week 216: number analyzed (Participants) | 0 | 37
  Week 216 |  | 73.70

5. Secondary Outcome: Annualized Relapse Rate (ARR) During the DB Period
Description: The ARR is calculated as the total number of participants with relapses experienced divided by the patient-years at risk. Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neurological NMO or NMOSD. Symptoms had to persist for >24 hours and not be attributable to confounding clinical factors (e.g., fever, infection, injury, change in mood, adverse reactions to medications). New or worsening neurological symptoms that occurred < 31 days following onset of a protocol-defined relapse were considered part of same relapse (2 relapses with onset days in 30 days of one another was counted as 1 relapse), onset date used in analysis was the date of first relapse.
Time Frame: Up to Week 216
Population: ITT population included all participants randomized to the treatment groups.
Measure: Number (95% Confidence Interval); unit: patients w relapse/patient-years at risk
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
patients w relapse/patient-years at risk | 0.32 [0.19 to 0.51] | 0.11 [0.05 to 0.21]

6. Secondary Outcome: Change From Baseline in Modified Rankin Scale (mRS) Scores at 24 Week Intervals During the DB Period
Description: The mRS is a 7-point disability scale that assesses the degree of disability in participants with neurological impairment. Possible scores range from 0 (no symptoms at all) up to 6 (death). Higher scores reflect increased disability. A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: ITT population included all participants randomized to the treatment groups. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 1.55 (0.97) | 1.90 (1.14)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | -0.03 (0.42) | -0.03 (0.50)
  Change from Baseline at Week 48: number analyzed (Participants) | 17 | 24
  Change from Baseline at Week 48 | -0.18 (0.53) | -0.13 (0.45)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 0.07 (0.70) | 0.00 (0.52)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 0.13 (0.62) | -0.19 (0.51)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | -0.10 (0.74) | -0.05 (0.51)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | -0.11 (0.93) | -0.20 (0.41)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | -0.67 (0.58) | -0.11 (0.33)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | -0.50 (0.71)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 0.00 (NA) — Standard deviation (SD) was not calculable for 1 participant.

7. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI) Scores at 24 Week Intervals During the DB Period
Description: The ZBI is the measurement to assess caregiver burden. The 22 items ask for the strain caregivers perceive. Responses range from 0 (never) to 4 (nearly always). The overall ZBI score ranges from 0 to 88. The higher the total score, the heavier the perceived burden. A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 168
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 16 | 13
score on scale
  Baseline | 19.31 (9.31) | 18.92 (12.82)
  Change from Baseline at Week 24: number analyzed (Participants) | 9 | 7
  Change from Baseline at Week 24 | -3.44 (5.59) | -3.57 (7.11)
  Change from Baseline at Week 48: number analyzed (Participants) | 6 | 8
  Change from Baseline at Week 48 | 1.17 (8.26) | 1.13 (13.45)
  Change from Baseline at Week 72: number analyzed (Participants) | 5 | 7
  Change from Baseline at Week 72 | 2.20 (19.64) | -0.71 (11.60)
  Change from Baseline at Week 96: number analyzed (Participants) | 5 | 6
  Change from Baseline at Week 96 | 3.00 (14.98) | 4.17 (13.33)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 5
  Change from Baseline at Week 120 | 0.00 (3.61) | 3.40 (9.29)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 4
  Change from Baseline at Week 144 | -3.50 (12.02) | -3.50 (11.33)
  Change from Baseline at Week 168: number analyzed (Participants) | 2 | 1
  Change from Baseline at Week 168 | 2.50 (13.44) | 11.00 (NA) — SD was not calculable for 1 participant.

8. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Scores at 24 Week Intervals During the DB Period
Description: The EDSS is an ordinal scale with values from 0 points (normal neurological examination) to 10 points (death) increasing in half-point increments once an EDSS of 1.0 has been reached. Higher scores represent increased disability. A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 41 | 41
score on scale
  Baseline | 3.63 (1.32) | 3.83 (1.57)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | -0.21 (0.68) | -0.14 (0.82)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | -0.19 (0.77) | -0.19 (0.67)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 21
  Change from Baseline at Week 72 | -0.27 (0.68) | -0.29 (0.73)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | -0.19 (0.81) | -0.19 (0.75)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | -0.30 (0.79) | 0.03 (0.57)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | -0.33 (0.83) | -0.07 (0.62)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | -0.17 (0.76) | -0.06 (0.58)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 0.00 (0.71)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | -0.50 (NA) — SD was not calculable for 1 participant.

9. Secondary Outcome: Change From Baseline in Visual Acuity (Snellen Chart) at 24 Week Intervals During the DB Period
Description: Visual acuity was measured using Snellen 20-foot wall chart and then converted to logMAR visual acuity scoring. Lower values indicate better visual acuity. Data are reported for right eye (OD) and left eye (OS). A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: LogMAR units
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
LogMAR units
  Baseline: OD | 0.490 (0.928) | 0.303 (0.593)
  Baseline: OS | 0.526 (0.911) | 0.597 (1.016)
  Change from Baseline at Week 24: OD: number analyzed (Participants) | 30 | 29
  Change from Baseline at Week 24: OD | -0.064 (0.197) | 0.042 (0.236)
  Change from Baseline at Week 24: OS: number analyzed (Participants) | 30 | 29
  Change from Baseline at Week 24: OS | -0.012 (0.107) | 0.059 (0.319)
  Change from Baseline at Week 48: OD: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48: OD | -0.019 (0.086) | 0.008 (0.093)
  Change from Baseline at Week 48: OS: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48: OS | 0.026 (0.096) | 0.013 (0.061)
  Change from Baseline at Week 72: OD: number analyzed (Participants) | 15 | 21
  Change from Baseline at Week 72: OD | -0.001 (0.110) | -0.034 (0.111)
  Change from Baseline at Week 72: OS: number analyzed (Participants) | 15 | 21
  Change from Baseline at Week 72: OS | -0.001 (0.121) | -0.019 (0.077)
  Change from Baseline at Week 96: OD: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96: OD | 0.018 (0.174) | -0.013 (0.095)
  Change from Baseline at Week 96: OS: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96: OS | -0.078 (0.185) | -0.010 (0.073)
  Change from Baseline at Week 120: OD: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120: OD | 0.030 (0.150) | 0.011 (0.103)
  Change from Baseline at Week 120: OS: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120: OS | -0.024 (0.150) | 0.014 (0.257)
  Change from Baseline at Week 144: OD: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144: OD | 0.058 (0.231) | -0.016 (0.120)
  Change from Baseline at Week 144: OS: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144: OS | -0.016 (0.165) | -0.028 (0.111)
  Change from Baseline at Week 168: OD: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168: OD | 0.113 (0.306) | 0.027 (0.199)
  Change from Baseline at Week 168: OS: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168: OS | 0.100 (0.173) | -0.024 (0.113)
  Change from Baseline at Week 192: OD: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192: OD |  | 0.150 (0.099)
  Change from Baseline at Week 192: OS: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192: OS |  | 0.000 (0.000)
  Change from Baseline at Week 216: OD: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216: OD |  | 0.120 (NA) — SD was not calculable for 1 participant.
  Change from Baseline at Week 216: OS: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216: OS |  | 0.000 (NA) — SD was not calculable for 1 participant.

10. Secondary Outcome: Change From Baseline in Short Form Generic Health Survey (SF-36) Mental Component Summary Scores at 24 Week Intervals During the DB Period
Description: The SF-36v2 is a multi-purpose, short form health survey with 36 questions. It has 8 domains (vitality, physical functioning, bodily pain, general health, role-physical, role emotional, social role functioning and mental health) of functional health and well-being scores as well as psychometrically based physical and mental health summary measures and a preference-based health utility index. The component scores were transformed to a 0-100 scale, where higher score indicates better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 44.77 (11.08) | 44.56 (9.75)
  Change from Baseline at Week 24: number analyzed (Participants) | 28 | 29
  Change from Baseline at Week 24 | 2.53 (7.58) | 0.57 (8.99)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 2.78 (7.51) | -0.61 (10.97)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 3.47 (7.13) | 2.78 (8.13)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 5.16 (10.52) | 1.06 (7.63)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 3.63 (8.62) | 0.71 (7.23)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 2.83 (8.79) | 3.82 (7.15)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 2.79 (6.85) | 3.60 (9.50)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 11.60 (7.32)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 14.05 (NA) — SD was not calculable for 1 participant.

11. Secondary Outcome: Change From Baseline in SF-36 Physical Component Summary Scores at 24 Week Intervals During the DB Period
Description: as for outcome 10
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 41.54 (9.11) | 43.60 (10.47)
  Change from Baseline at Week 24: number analyzed (Participants) | 28 | 29
  Change from Baseline at Week 24 | 2.79 (5.61) | 1.30 (6.01)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 0.18 (5.33) | 1.22 (5.77)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 1.97 (6.23) | 1.16 (4.79)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | -1.15 (7.52) | 1.88 (5.72)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | -0.13 (7.10) | 2.34 (6.60)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 1.78 (5.50) | 3.05 (4.23)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 0.22 (9.23) | 0.76 (5.98)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 0.23 (0.55)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | -1.63 (NA) — SD was not calculable for 1 participant.

12. Secondary Outcome: Change From Baseline in SF-36 Bodily Pain Domain Scores at 24 Week Intervals During the DB Period
Description: The SF-36v2 is a multi-purpose, short form health survey with 36 questions. It has 8 domains (vitality, physical functioning, bodily pain, general health, role-physical, role emotional, social role functioning and mental health) of functional health and well-being scores as well as psychometrically based physical and mental health component summary measures and a preference-based health utility index. The domain scores were transformed to a 0-100 scale, where higher scores indicate better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 43.91 (10.22) | 45.94 (11.56)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | 2.71 (7.06) | 0.03 (11.06)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 0.81 (5.60) | 0.12 (6.99)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 3.55 (8.20) | 2.30 (6.99)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 1.31 (7.13) | 1.15 (8.86)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 2.22 (9.96) | -1.45 (9.13)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 3.58 (8.53) | 3.14 (8.18)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 1.61 (10.58) | 3.05 (9.00)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 8.07 (0.57)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 3.63 (NA) — SD was not calculable for 1 participant.

13. Secondary Outcome: Change From Baseline in SF-36 General Health Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 39.65 (7.90) | 41.23 (9.29)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | 1.84 (5.68) | -0.60 (7.26)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | -0.66 (5.53) | -0.27 (6.00)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | -0.16 (6.25) | 0.94 (5.57)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | -1.90 (6.17) | 1.86 (6.12)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | -0.33 (4.03) | 3.76 (6.72)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | -0.95 (5.66) | 5.20 (7.11)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | -5.23 (7.41) | 3.06 (6.99)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 1.19 (5.04)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | -2.38 (NA) — SD was not calculable for 1 participant.

14. Secondary Outcome: Change From Baseline in SF-36 Mental Health Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 43.71 (10.92) | 43.59 (10.55)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | 5.23 (7.69) | 0.99 (10.21)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 2.76 (8.54) | 0.11 (10.73)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 5.23 (7.66) | 3.18 (9.72)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 4.09 (8.49) | 2.12 (8.13)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 3.14 (7.06) | 1.57 (6.76)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 3.49 (7.04) | 4.88 (8.38)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 4.36 (3.02) | 4.07 (10.72)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 13.09 (14.80)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 23.55 (NA) — SD was not calculable for 1 participant.

15. Secondary Outcome: Change From Baseline in SF-36 Physical Functioning Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 42.50 (10.53) | 43.46 (10.34)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | 3.56 (7.04) | 1.49 (7.05)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 1.92 (4.30) | 1.86 (7.73)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 3.19 (6.54) | 0.88 (6.52)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 0.84 (6.77) | 2.37 (7.75)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | -0.19 (8.39) | 2.58 (6.03)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 2.55 (4.06) | 3.32 (5.72)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 1.92 (5.06) | 0.00 (5.50)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 1.91 (2.70)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 1.91 (NA) — SD was not calculable for 1 participant.

16. Secondary Outcome: Change From Baseline in SF-36 Role-Emotional Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 43.98 (11.46) | 43.01 (10.55)
  Change from Baseline at Week 24: number analyzed (Participants) | 28 | 29
  Change from Baseline at Week 24 | 2.24 (10.35) | 0.36 (10.12)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 3.29 (8.05) | 0.00 (12.49)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 1.39 (9.38) | 2.57 (7.66)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 4.13 (14.40) | 0.83 (10.20)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 3.13 (12.44) | 0.35 (6.95)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 3.09 (9.61) | 3.25 (7.38)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 1.16 (5.32) | 4.64 (9.05)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 12.19 (2.46)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 6.97 (NA) — SD was not calculable for 1 participant.

17. Secondary Outcome: Change From Baseline in SF-36 Role-Physical Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 40.74 (10.12) | 41.88 (11.38)
  Change from Baseline at Week 24: number analyzed (Participants) | 28 | 29
  Change from Baseline at Week 24 | 3.93 (9.56) | 3.02 (6.95)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 1.37 (7.23) | 1.40 (8.66)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 2.40 (7.94) | 2.83 (7.81)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 0.42 (9.03) | 1.71 (4.60)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 1.57 (9.47) | 3.14 (7.44)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 2.99 (6.05) | 2.69 (6.80)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 3.74 (10.61) | 2.25 (6.45)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 4.49 (6.35)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 8.98 (NA) — SD was not calculable for 1 participant.

18. Secondary Outcome: Change From Baseline in SF-36 Social Role Functioning Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 41.70 (11.62) | 44.26 (10.92)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | 1.73 (7.96) | 0.86 (8.69)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 1.12 (7.80) | 0.00 (10.24)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 2.34 (7.78) | 2.18 (7.22)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 2.82 (11.72) | 0.00 (9.38)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 1.51 (13.59) | 0.25 (9.13)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 0.56 (9.85) | 2.01 (7.29)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 1.67 (22.61) | 0.00 (5.61)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 0.00 (0.00)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | -5.01 (NA) — SD was not calculable for 1 participant.

19. Secondary Outcome: Change From Baseline in SF-36 Vitality Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 12
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
score on scale
  Baseline | 45.95 (9.14) | 46.66 (9.65)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 29
  Change from Baseline at Week 24 | 2.66 (7.38) | 1.74 (8.61)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 24
  Change from Baseline at Week 48 | 1.65 (5.60) | -0.25 (8.71)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 23
  Change from Baseline at Week 72 | 4.55 (6.91) | 1.38 (9.12)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 21
  Change from Baseline at Week 96 | 4.08 (8.53) | 2.41 (8.28)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 20
  Change from Baseline at Week 120 | 2.97 (5.24) | 2.67 (8.45)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 3.96 (6.12) | 4.16 (10.03)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 2.97 (2.97) | 0.99 (10.82)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 7.43 (10.51)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 11.89 (NA) — SD was not calculable for 1 participant.

20. Secondary Outcome: Change From Baseline in EuroQoL-5 Dimensions (EQ-5D) Index Scores at 24 Week Intervals During the DB Period
Description: The EQ-5D is a participant-answered questionnaire measuring 5 dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with 3 possible response categories: 1) no problems; 2) some problems; 3) severe problems. The scores from 5 dimensions are used as input to generate EQ-5D index score using scoring algorithm. The EQ-5D index score is scored on a scale of -0.2 to 1. A higher score reflects a better health state. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 40
score on scale
  Baseline | 0.7297 (0.1863) | 0.7634 (0.1811)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 28
  Change from Baseline at Week 24 | 0.0649 (0.1596) | -0.0082 (0.1882)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 23
  Change from Baseline at Week 48 | 0.0352 (0.1830) | 0.0011 (0.1256)
  Change from Baseline at Week 72: number analyzed (Participants) | 15 | 22
  Change from Baseline at Week 72 | 0.0724 (0.2088) | 0.0241 (0.1084)
  Change from Baseline at Week 96: number analyzed (Participants) | 16 | 20
  Change from Baseline at Week 96 | 0.0349 (0.1758) | 0.0167 (0.1056)
  Change from Baseline at Week 120: number analyzed (Participants) | 10 | 19
  Change from Baseline at Week 120 | 0.0336 (0.2111) | 0.0257 (0.1178)
  Change from Baseline at Week 144: number analyzed (Participants) | 9 | 15
  Change from Baseline at Week 144 | 0.0846 (0.1650) | 0.0488 (0.1424)
  Change from Baseline at Week 168: number analyzed (Participants) | 3 | 9
  Change from Baseline at Week 168 | 0.0648 (0.1031) | 0.0307 (0.1335)
  Change from Baseline at Week 192: number analyzed (Participants) | 0 | 2
  Change from Baseline at Week 192 |  | 0.1873 (0.2890)
  Change from Baseline at Week 216: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 216 |  | 0.3322 (NA) — SD was not calculable for 1 participant.

21. Secondary Outcome: Serum Satralizumab Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, 5, 6, 8, and every 4 weeks thereafter up to Week 224
Population: Participants from Safety Analysis Population (SAF) who received satralizumab were evaluated for this outcome measure. The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 41
ng/mL
  Baseline: number analyzed (Participants) | 40
  Baseline | 100.00 (0.00)
  Week 2 | 11343.66 (5125.84)
  Week 4: number analyzed (Participants) | 38
  Week 4 | 22222.63 (8003.48)
  Week 5: number analyzed (Participants) | 20
  Week 5 | 28461.00 (12542.52)
  Week 6: number analyzed (Participants) | 20
  Week 6 | 28174.50 (11199.00)
  Week 8: number analyzed (Participants) | 39
  Week 8 | 21246.92 (9045.31)
  Week 12: number analyzed (Participants) | 38
  Week 12 | 20927.63 (9536.07)
  Week 16: number analyzed (Participants) | 35
  Week 16 | 20274.86 (10694.38)
  Week 20: number analyzed (Participants) | 33
  Week 20 | 20146.06 (10740.65)
  Week 24: number analyzed (Participants) | 30
  Week 24 | 20189.00 (10140.88)
  Week 28: number analyzed (Participants) | 28
  Week 28 | 20826.07 (10995.92)
  Week 32: number analyzed (Participants) | 28
  Week 32 | 20631.79 (11110.94)
  Week 36: number analyzed (Participants) | 26
  Week 36 | 21114.62 (11190.52)
  Week 40: number analyzed (Participants) | 25
  Week 40 | 22224.76 (13389.71)
  Week 44: number analyzed (Participants) | 23
  Week 44 | 22582.17 (12031.13)
  Week 48: number analyzed (Participants) | 25
  Week 48 | 23324.80 (13979.87)
  Week 52: number analyzed (Participants) | 24
  Week 52 | 24570.83 (15798.38)
  Week 56: number analyzed (Participants) | 24
  Week 56 | 24252.50 (15433.80)
  Week 60: number analyzed (Participants) | 24
  Week 60 | 23061.67 (15777.82)
  Week 64: number analyzed (Participants) | 22
  Week 64 | 23369.55 (13447.96)
  Week 68: number analyzed (Participants) | 23
  Week 68 | 26194.43 (16836.77)
  Week 72: number analyzed (Participants) | 23
  Week 72 | 26618.87 (14999.38)
  Week 76: number analyzed (Participants) | 22
  Week 76 | 26539.09 (13736.30)
  Week 80: number analyzed (Participants) | 21
  Week 80 | 26868.00 (14005.87)
  Week 84: number analyzed (Participants) | 21
  Week 84 | 27037.62 (15460.97)
  Week 88: number analyzed (Participants) | 20
  Week 88 | 26203.00 (14309.81)
  Week 92: number analyzed (Participants) | 21
  Week 92 | 28308.10 (15111.34)
  Week 96: number analyzed (Participants) | 21
  Week 96 | 26754.43 (15146.20)
  Week 100: number analyzed (Participants) | 21
  Week 100 | 27707.14 (14225.93)
  Week 104: number analyzed (Participants) | 21
  Week 104 | 26203.81 (13616.28)
  Week 108: number analyzed (Participants) | 21
  Week 108 | 26112.38 (12521.65)
  Week 112: number analyzed (Participants) | 21
  Week 112 | 24925.10 (12181.81)
  Week 116: number analyzed (Participants) | 20
  Week 116 | 26360.50 (13885.76)
  Week 120: number analyzed (Participants) | 20
  Week 120 | 24910.00 (13217.57)
  Week 124: number analyzed (Participants) | 20
  Week 124 | 24689.50 (14352.30)
  Week 128: number analyzed (Participants) | 19
  Week 128 | 22395.53 (12954.00)
  Week 132: number analyzed (Participants) | 19
  Week 132 | 23804.74 (14878.32)
  Week 136: number analyzed (Participants) | 19
  Week 136 | 25856.32 (15506.85)
  Week 140: number analyzed (Participants) | 18
  Week 140 | 26118.56 (15264.89)
  Week 144: number analyzed (Participants) | 15
  Week 144 | 27975.33 (11536.28)
  Week 148: number analyzed (Participants) | 12
  Week 148 | 27935.83 (11940.90)
  Week 152: number analyzed (Participants) | 10
  Week 152 | 28967.00 (10354.22)
  Week 156: number analyzed (Participants) | 9
  Week 156 | 27990.00 (10444.75)
  Week 160: number analyzed (Participants) | 9
  Week 160 | 28983.33 (11429.02)
  Week 164: number analyzed (Participants) | 9
  Week 164 | 28903.33 (10780.69)
  Week 168: number analyzed (Participants) | 9
  Week 168 | 23683.33 (11615.40)
  Week 172: number analyzed (Participants) | 9
  Week 172 | 24498.89 (11106.23)
  Week 176: number analyzed (Participants) | 9
  Week 176 | 26300.00 (11498.48)
  Week 180: number analyzed (Participants) | 6
  Week 180 | 28300.00 (9431.86)
  Week 184: number analyzed (Participants) | 5
  Week 184 | 32380.00 (9427.19)
  Week 188: number analyzed (Participants) | 3
  Week 188 | 36600.00 (8214.62)
  Week 192: number analyzed (Participants) | 2
  Week 192 | 32650.00 (7848.89)
  Week 196: number analyzed (Participants) | 2
  Week 196 | 30800.00 (4808.33)
  Week 200: number analyzed (Participants) | 2
  Week 200 | 28400.00 (3818.38)
  Week 204: number analyzed (Participants) | 2
  Week 204 | 25300.00 (3252.69)
  Week 208: number analyzed (Participants) | 1
  Week 208 | 25900.00 (NA) — SD was not calculable for 1 participant.
  Week 212: number analyzed (Participants) | 1
  Week 212 | 17000.00 (NA) — SD was not calculable for 1 participant.
  Week 216: number analyzed (Participants) | 1
  Week 216 | 28600.00 (NA) — SD was not calculable for 1 participant.
  Week 220: number analyzed (Participants) | 1
  Week 220 | 31600.00 (NA) — SD was not calculable for 1 participant.
  Week 224: number analyzed (Participants) | 1
  Week 224 | 28700.00 (NA) — SD was not calculable for 1 participant.

22. Secondary Outcome: Serum Soluble IL-6 Receptor (sIL-6R) Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, and every 4 weeks thereafter up to Week 224
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
ng/mL
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 32.52 (7.78) | 35.13 (21.52)
  Week 2: number analyzed (Participants) | 41 | 41
  Week 2 | 33.82 (8.30) | 437.41 (72.31)
  Week 4: number analyzed (Participants) | 40 | 41
  Week 4 | 33.13 (8.52) | 572.29 (94.84)
  Week 8: number analyzed (Participants) | 37 | 39
  Week 8 | 34.02 (9.43) | 642.92 (115.51)
  Week 12: number analyzed (Participants) | 33 | 39
  Week 12 | 32.58 (8.52) | 651.41 (99.20)
  Week 16: number analyzed (Participants) | 32 | 35
  Week 16 | 32.67 (9.32) | 640.57 (97.41)
  Week 20: number analyzed (Participants) | 31 | 33
  Week 20 | 34.22 (8.15) | 636.64 (109.75)
  Week 24: number analyzed (Participants) | 30 | 30
  Week 24 | 34.44 (9.31) | 639.20 (108.94)
  Week 28: number analyzed (Participants) | 26 | 28
  Week 28 | 33.70 (8.28) | 649.11 (131.85)
  Week 32: number analyzed (Participants) | 24 | 28
  Week 32 | 33.48 (8.74) | 651.82 (162.04)
  Week 36: number analyzed (Participants) | 23 | 26
  Week 36 | 34.39 (11.01) | 652.12 (124.70)
  Week 40: number analyzed (Participants) | 19 | 24
  Week 40 | 33.31 (7.86) | 664.21 (158.61)
  Week 44: number analyzed (Participants) | 18 | 23
  Week 44 | 33.94 (7.77) | 677.13 (173.99)
  Week 48: number analyzed (Participants) | 18 | 25
  Week 48 | 34.50 (9.14) | 627.23 (217.06)
  Week 52: number analyzed (Participants) | 18 | 24
  Week 52 | 44.01 (44.26) | 656.29 (173.67)
  Week 56: number analyzed (Participants) | 18 | 24
  Week 56 | 37.00 (7.42) | 626.83 (155.56)
  Week 60: number analyzed (Participants) | 18 | 24
  Week 60 | 36.39 (7.81) | 617.00 (142.13)
  Week 64: number analyzed (Participants) | 17 | 22
  Week 64 | 35.14 (8.78) | 621.27 (152.45)
  Week 68: number analyzed (Participants) | 17 | 23
  Week 68 | 35.35 (8.68) | 664.91 (130.58)
  Week 72: number analyzed (Participants) | 15 | 23
  Week 72 | 36.02 (10.73) | 648.83 (134.32)
  Week 76: number analyzed (Participants) | 16 | 22
  Week 76 | 36.94 (9.46) | 643.91 (118.60)
  Week 80: number analyzed (Participants) | 16 | 21
  Week 80 | 36.45 (9.50) | 667.24 (133.49)
  Week 84: number analyzed (Participants) | 16 | 21
  Week 84 | 34.60 (8.88) | 649.38 (137.64)
  Week 88: number analyzed (Participants) | 13 | 20
  Week 88 | 31.95 (8.29) | 651.35 (150.58)
  Week 92: number analyzed (Participants) | 16 | 21
  Week 92 | 34.30 (9.71) | 633.43 (134.36)
  Week 96: number analyzed (Participants) | 16 | 21
  Week 96 | 32.88 (9.39) | 630.62 (162.28)
  Week 100: number analyzed (Participants) | 15 | 21
  Week 100 | 33.78 (9.04) | 651.90 (162.09)
  Week 104: number analyzed (Participants) | 14 | 21
  Week 104 | 31.61 (9.13) | 649.57 (185.99)
  Week 108: number analyzed (Participants) | 13 | 21
  Week 108 | 31.49 (9.23) | 658.67 (152.61)
  Week 112: number analyzed (Participants) | 12 | 21
  Week 112 | 32.75 (7.77) | 683.90 (135.07)
  Week 116: number analyzed (Participants) | 13 | 20
  Week 116 | 33.68 (8.31) | 653.98 (194.92)
  Week 120: number analyzed (Participants) | 12 | 20
  Week 120 | 33.73 (6.20) | 667.10 (152.24)
  Week 124: number analyzed (Participants) | 10 | 20
  Week 124 | 33.06 (9.31) | 696.45 (138.17)
  Week 128: number analyzed (Participants) | 10 | 19
  Week 128 | 34.07 (8.83) | 670.05 (138.28)
  Week 132: number analyzed (Participants) | 10 | 19
  Week 132 | 34.28 (4.95) | 671.84 (138.75)
  Week 136: number analyzed (Participants) | 10 | 19
  Week 136 | 32.43 (8.12) | 674.95 (170.04)
  Week 140: number analyzed (Participants) | 10 | 18
  Week 140 | 32.97 (6.52) | 645.72 (132.32)
  Week 144: number analyzed (Participants) | 9 | 15
  Week 144 | 35.37 (8.91) | 699.80 (101.84)
  Week 148: number analyzed (Participants) | 7 | 12
  Week 148 | 37.97 (12.40) | 672.42 (107.40)
  Week 152: number analyzed (Participants) | 5 | 10
  Week 152 | 35.08 (9.08) | 701.60 (110.27)
  Week 156: number analyzed (Participants) | 5 | 9
  Week 156 | 36.92 (7.77) | 720.33 (103.58)
  Week 160: number analyzed (Participants) | 4 | 9
  Week 160 | 40.38 (7.31) | 704.89 (109.86)
  Week 164: number analyzed (Participants) | 4 | 9
  Week 164 | 43.08 (10.54) | 723.67 (136.20)
  Week 168: number analyzed (Participants) | 3 | 9
  Week 168 | 42.30 (5.92) | 744.22 (123.47)
  Week 172: number analyzed (Participants) | 3 | 9
  Week 172 | 42.03 (5.87) | 706.33 (127.63)
  Week 176: number analyzed (Participants) | 2 | 9
  Week 176 | 39.85 (6.15) | 730.56 (121.75)
  Week 180: number analyzed (Participants) | 2 | 6
  Week 180 | 38.85 (12.09) | 769.83 (119.50)
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 736.80 (152.09)
  Week 188: number analyzed (Participants) | 0 | 3
  Week 188 |  | 853.67 (38.02)
  Week 192: number analyzed (Participants) | 0 | 2
  Week 192 |  | 930.00 (49.50)
  Week 196: number analyzed (Participants) | 0 | 2
  Week 196 |  | 887.00 (91.92)
  Week 200: number analyzed (Participants) | 0 | 2
  Week 200 |  | 902.50 (79.90)
  Week 204: number analyzed (Participants) | 0 | 2
  Week 204 |  | 935.00 (7.07)
  Week 208: number analyzed (Participants) | 0 | 1
  Week 208 |  | 941.00 (NA) — SD was not calculable for 1 participant.
  Week 212: number analyzed (Participants) | 0 | 1
  Week 212 |  | 971.00 (NA) — SD was not calculable for 1 participant.
  Week 216: number analyzed (Participants) | 0 | 1
  Week 216 |  | 896.00 (NA) — SD was not calculable for 1 participant.
  Week 220: number analyzed (Participants) | 0 | 1
  Week 220 |  | 901.00 (NA) — SD was not calculable for 1 participant.
  Week 224: number analyzed (Participants) | 0 | 1
  Week 224 |  | 831.00 (NA) — SD was not calculable for 1 participant.

23. Secondary Outcome: Serum High Sensitivity C-Reactive Protein (hsCRP) Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, and every 4 weeks thereafter up to Week 224
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
mg/L
  Baseline | 1.48 (2.08) | 1.68 (2.49)
  Week 2: number analyzed (Participants) | 41 | 40
  Week 2 | 1.65 (2.86) | 0.78 (2.93)
  Week 4: number analyzed (Participants) | 40 | 41
  Week 4 | 1.59 (2.27) | 0.44 (0.72)
  Week 8: number analyzed (Participants) | 37 | 39
  Week 8 | 1.76 (2.25) | 0.59 (1.26)
  Week 12: number analyzed (Participants) | 33 | 38
  Week 12 | 1.48 (2.07) | 0.47 (0.60)
  Week 16: number analyzed (Participants) | 32 | 35
  Week 16 | 1.91 (3.34) | 0.49 (0.51)
  Week 20: number analyzed (Participants) | 31 | 33
  Week 20 | 1.91 (3.44) | 0.48 (0.50)
  Week 24: number analyzed (Participants) | 30 | 30
  Week 24 | 2.45 (6.87) | 0.58 (0.91)
  Week 28: number analyzed (Participants) | 26 | 28
  Week 28 | 1.96 (3.24) | 0.73 (1.34)
  Week 32: number analyzed (Participants) | 24 | 28
  Week 32 | 2.36 (4.96) | 0.73 (1.21)
  Week 36: number analyzed (Participants) | 23 | 26
  Week 36 | 2.48 (3.59) | 0.56 (0.66)
  Week 40: number analyzed (Participants) | 19 | 25
  Week 40 | 2.49 (4.53) | 1.13 (2.26)
  Week 44: number analyzed (Participants) | 18 | 23
  Week 44 | 1.41 (1.47) | 0.72 (1.20)
  Week 48: number analyzed (Participants) | 18 | 25
  Week 48 | 1.59 (2.07) | 0.86 (1.44)
  Week 52: number analyzed (Participants) | 18 | 24
  Week 52 | 2.60 (3.87) | 0.67 (0.88)
  Week 56: number analyzed (Participants) | 18 | 23
  Week 56 | 1.43 (1.58) | 0.72 (1.02)
  Week 60: number analyzed (Participants) | 18 | 24
  Week 60 | 2.63 (4.34) | 1.05 (2.15)
  Week 64: number analyzed (Participants) | 17 | 22
  Week 64 | 11.10 (40.09) | 0.64 (0.89)
  Week 68: number analyzed (Participants) | 17 | 23
  Week 68 | 1.86 (2.66) | 0.57 (0.47)
  Week 72: number analyzed (Participants) | 15 | 23
  Week 72 | 3.80 (8.83) | 0.59 (0.71)
  Week 76: number analyzed (Participants) | 15 | 22
  Week 76 | 5.24 (10.68) | 0.51 (0.37)
  Week 80: number analyzed (Participants) | 16 | 21
  Week 80 | 2.11 (2.63) | 0.58 (0.51)
  Week 84: number analyzed (Participants) | 16 | 21
  Week 84 | 2.08 (2.26) | 0.59 (0.61)
  Week 88: number analyzed (Participants) | 14 | 20
  Week 88 | 5.19 (12.83) | 0.60 (0.53)
  Week 92: number analyzed (Participants) | 16 | 21
  Week 92 | 2.07 (2.21) | 0.60 (0.70)
  Week 96: number analyzed (Participants) | 16 | 20
  Week 96 | 2.92 (4.60) | 0.74 (1.01)
  Week 100: number analyzed (Participants) | 15 | 21
  Week 100 | 2.58 (4.53) | 0.87 (1.49)
  Week 104: number analyzed (Participants) | 14 | 21
  Week 104 | 1.41 (2.05) | 0.84 (1.40)
  Week 108: number analyzed (Participants) | 13 | 21
  Week 108 | 1.93 (2.25) | 0.66 (0.58)
  Week 112: number analyzed (Participants) | 12 | 21
  Week 112 | 1.54 (1.56) | 0.82 (0.87)
  Week 116: number analyzed (Participants) | 13 | 20
  Week 116 | 2.39 (3.91) | 0.84 (1.26)
  Week 120: number analyzed (Participants) | 12 | 20
  Week 120 | 1.53 (1.33) | 0.98 (1.58)
  Week 124: number analyzed (Participants) | 10 | 20
  Week 124 | 1.43 (1.43) | 0.72 (0.67)
  Week 128: number analyzed (Participants) | 10 | 19
  Week 128 | 6.00 (16.28) | 0.96 (1.29)
  Week 132: number analyzed (Participants) | 10 | 19
  Week 132 | 1.08 (0.94) | 0.70 (0.84)
  Week 136: number analyzed (Participants) | 10 | 19
  Week 136 | 1.43 (1.54) | 0.99 (1.68)
  Week 140: number analyzed (Participants) | 10 | 18
  Week 140 | 1.15 (1.28) | 1.06 (2.25)
  Week 144: number analyzed (Participants) | 9 | 15
  Week 144 | 0.82 (0.73) | 0.44 (0.37)
  Week 148: number analyzed (Participants) | 7 | 12
  Week 148 | 1.29 (1.43) | 0.35 (0.18)
  Week 152: number analyzed (Participants) | 5 | 10
  Week 152 | 1.08 (0.97) | 0.38 (0.23)
  Week 156: number analyzed (Participants) | 5 | 9
  Week 156 | 1.52 (1.42) | 0.35 (0.18)
  Week 160: number analyzed (Participants) | 4 | 9
  Week 160 | 0.83 (0.53) | 0.37 (0.22)
  Week 164: number analyzed (Participants) | 4 | 9
  Week 164 | 3.18 (4.89) | 0.38 (0.20)
  Week 168: number analyzed (Participants) | 3 | 9
  Week 168 | 0.80 (0.26) | 0.40 (0.19)
  Week 172: number analyzed (Participants) | 3 | 8
  Week 172 | 1.37 (1.00) | 0.26 (0.17)
  Week 176: number analyzed (Participants) | 2 | 8
  Week 176 | 0.95 (0.64) | 0.31 (0.19)
  Week 180: number analyzed (Participants) | 2 | 6
  Week 180 | 30.15 (41.65) | 0.28 (0.15)
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 0.20 (0.11)
  Week 188: number analyzed (Participants) | 0 | 3
  Week 188 |  | 0.37 (0.06)
  Week 192: number analyzed (Participants) | 0 | 2
  Week 192 |  | 0.15 (0.00)
  Week 196: number analyzed (Participants) | 0 | 2
  Week 196 |  | 0.23 (0.11)
  Week 200: number analyzed (Participants) | 0 | 2
  Week 200 |  | 0.23 (0.11)
  Week 204: number analyzed (Participants) | 0 | 2
  Week 204 |  | 0.23 (0.11)
  Week 208: number analyzed (Participants) | 0 | 1
  Week 208 |  | 0.30 (NA) — SD was not calculable for 1 participant.
  Week 212: number analyzed (Participants) | 0 | 1
  Week 212 |  | 0.40 (NA) — SD was not calculable for 1 participant.
  Week 216: number analyzed (Participants) | 0 | 1
  Week 216 |  | 0.30 (NA) — SD was not calculable for 1 participant.
  Week 220: number analyzed (Participants) | 0 | 1
  Week 220 |  | 0.40 (NA) — SD was not calculable for 1 participant.
  Week 224: number analyzed (Participants) | 0 | 1
  Week 224 |  | 0.15 (NA) — SD was not calculable for 1 participant.

24. Secondary Outcome: Serum Interleukin-6 (IL-6) Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, and every 4 weeks thereafter up to Week 224
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
pg/mL
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 1.63 (0.39) | 1.92 (1.36)
  Week 2: number analyzed (Participants) | 41 | 41
  Week 2 | 1.84 (0.95) | 40.12 (118.83)
  Week 4: number analyzed (Participants) | 40 | 41
  Week 4 | 2.33 (2.99) | 28.30 (31.31)
  Week 8: number analyzed (Participants) | 37 | 38
  Week 8 | 1.69 (0.55) | 32.37 (77.99)
  Week 12: number analyzed (Participants) | 33 | 39
  Week 12 | 1.71 (0.60) | 22.95 (20.55)
  Week 16: number analyzed (Participants) | 32 | 35
  Week 16 | 1.84 (0.90) | 25.76 (30.85)
  Week 20: number analyzed (Participants) | 31 | 33
  Week 20 | 2.99 (5.45) | 23.07 (15.37)
  Week 24: number analyzed (Participants) | 30 | 29
  Week 24 | 2.02 (1.52) | 21.53 (17.91)
  Week 28: number analyzed (Participants) | 26 | 28
  Week 28 | 1.95 (1.38) | 25.14 (24.27)
  Week 32: number analyzed (Participants) | 24 | 28
  Week 32 | 1.74 (0.84) | 23.77 (18.53)
  Week 36: number analyzed (Participants) | 23 | 26
  Week 36 | 2.13 (1.41) | 23.08 (15.56)
  Week 40: number analyzed (Participants) | 19 | 24
  Week 40 | 1.66 (0.40) | 27.31 (47.45)
  Week 44: number analyzed (Participants) | 17 | 21
  Week 44 | 1.57 (0.00) | 17.01 (15.38)
  Week 48: number analyzed (Participants) | 18 | 25
  Week 48 | 1.69 (0.53) | 19.45 (19.36)
  Week 52: number analyzed (Participants) | 18 | 24
  Week 52 | 2.12 (1.36) | 21.11 (17.42)
  Week 56: number analyzed (Participants) | 18 | 22
  Week 56 | 1.57 (0.00) | 21.74 (20.96)
  Week 60: number analyzed (Participants) | 18 | 23
  Week 60 | 2.27 (1.46) | 23.25 (23.36)
  Week 64: number analyzed (Participants) | 17 | 22
  Week 64 | 2.46 (3.22) | 24.31 (20.74)
  Week 68: number analyzed (Participants) | 17 | 23
  Week 68 | 1.94 (1.14) | 31.30 (53.79)
  Week 72: number analyzed (Participants) | 15 | 23
  Week 72 | 1.93 (0.97) | 24.69 (24.45)
  Week 76: number analyzed (Participants) | 16 | 21
  Week 76 | 2.21 (1.87) | 20.45 (13.79)
  Week 80: number analyzed (Participants) | 16 | 21
  Week 80 | 2.19 (2.51) | 23.29 (19.64)
  Week 84: number analyzed (Participants) | 16 | 21
  Week 84 | 2.66 (2.36) | 22.71 (21.49)
  Week 88: number analyzed (Participants) | 12 | 20
  Week 88 | 2.59 (2.77) | 29.17 (25.58)
  Week 92: number analyzed (Participants) | 16 | 20
  Week 92 | 1.84 (0.77) | 24.51 (32.02)
  Week 96: number analyzed (Participants) | 16 | 21
  Week 96 | 3.06 (3.19) | 21.52 (20.20)
  Week 100: number analyzed (Participants) | 15 | 21
  Week 100 | 2.04 (1.02) | 21.77 (24.98)
  Week 104: number analyzed (Participants) | 13 | 21
  Week 104 | 1.95 (0.96) | 22.61 (26.55)
  Week 108: number analyzed (Participants) | 13 | 21
  Week 108 | 1.76 (0.70) | 24.18 (20.55)
  Week 112: number analyzed (Participants) | 12 | 21
  Week 112 | 1.57 (0.00) | 32.18 (36.15)
  Week 116: number analyzed (Participants) | 13 | 20
  Week 116 | 1.57 (0.00) | 22.33 (22.20)
  Week 120: number analyzed (Participants) | 12 | 20
  Week 120 | 1.71 (0.52) | 21.86 (24.54)
  Week 124: number analyzed (Participants) | 9 | 19
  Week 124 | 1.57 (0.00) | 26.23 (27.67)
  Week 128: number analyzed (Participants) | 10 | 19
  Week 128 | 1.57 (0.00) | 25.40 (31.20)
  Week 132: number analyzed (Participants) | 10 | 19
  Week 132 | 1.57 (0.00) | 25.48 (27.38)
  Week 136: number analyzed (Participants) | 10 | 19
  Week 136 | 1.57 (0.00) | 27.23 (37.56)
  Week 140: number analyzed (Participants) | 10 | 18
  Week 140 | 1.57 (0.00) | 20.66 (18.10)
  Week 144: number analyzed (Participants) | 9 | 15
  Week 144 | 1.57 (0.00) | 16.82 (16.16)
  Week 148: number analyzed (Participants) | 7 | 12
  Week 148 | 2.04 (1.25) | 17.10 (11.33)
  Week 152: number analyzed (Participants) | 5 | 10
  Week 152 | 1.57 (0.00) | 16.62 (13.75)
  Week 156: number analyzed (Participants) | 5 | 8
  Week 156 | 2.34 (1.72) | 12.67 (5.73)
  Week 160: number analyzed (Participants) | 4 | 9
  Week 160 | 1.96 (0.80) | 11.15 (5.12)
  Week 164: number analyzed (Participants) | 4 | 9
  Week 164 | 1.57 (0.00) | 12.84 (6.93)
  Week 168: number analyzed (Participants) | 3 | 9
  Week 168 | 1.57 (0.00) | 13.30 (8.89)
  Week 172: number analyzed (Participants) | 3 | 9
  Week 172 | 1.57 (0.00) | 13.89 (6.94)
  Week 176: number analyzed (Participants) | 2 | 9
  Week 176 | 1.57 (0.00) | 15.11 (7.16)
  Week 180: number analyzed (Participants) | 2 | 6
  Week 180 | 1.57 (0.00) | 13.34 (6.68)
  Week 184: number analyzed (Participants) | 0 | 5
  Week 184 |  | 15.24 (9.91)
  Week 188: number analyzed (Participants) | 0 | 3
  Week 188 |  | 13.96 (9.74)
  Week 192: number analyzed (Participants) | 0 | 2
  Week 192 |  | 16.71 (13.15)
  Week 196: number analyzed (Participants) | 0 | 2
  Week 196 |  | 14.34 (12.81)
  Week 200: number analyzed (Participants) | 0 | 2
  Week 200 |  | 18.55 (8.84)
  Week 204: number analyzed (Participants) | 0 | 2
  Week 204 |  | 18.24 (12.53)
  Week 208: number analyzed (Participants) | 0 | 1
  Week 208 |  | 9.95 (NA) — SD was not calculable for 1 participant.
  Week 212: number analyzed (Participants) | 0 | 1
  Week 212 |  | 8.02 (NA) — SD was not calculable for 1 participant.
  Week 216: number analyzed (Participants) | 0 | 1
  Week 216 |  | 6.45 (NA) — SD was not calculable for 1 participant.
  Week 220: number analyzed (Participants) | 0 | 1
  Week 220 |  | 45.80 (NA) — SD was not calculable for 1 participant.
  Week 224: number analyzed (Participants) | 0 | 1
  Week 224 |  | 34.30 (NA) — SD was not calculable for 1 participant.

25. Secondary Outcome: Number of Participants With at Least One Adverse Event in the DB Period
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to Week 224
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
participants | 40 | 37

26. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event in the DB Period
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Week 224
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
participants | 9 | 7

27. Secondary Outcome: Number of Participants With Non-Serious Adverse Events of Special Interest in the DB Period
Description: Non-serious adverse events of special interest for this study included: 1) cases of an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice, 2) suspected transmission of an infectious agent by the study treatment.
Time Frame: Up to Week 224
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
participants | 0 | 0

28. Secondary Outcome: Number of Participants With Selected Adverse Events in the DB Period
Description: Selected adverse events for this study included: 1) non-serious infections that required treatments with intravenous (IV) antibiotic, antifungal, antiviral, 2) opportunistic infections that required treatments with oral antibiotics, antifungals, or antivirals, 3) injection-related reactions (IRRs; an AE which occured within 24 hours after study treatment injection except where the event was not considered an allergic reaction), and 4) anaphylaxis (an acute allergic/hypersensitivity reaction).
Time Frame: Up to Week 224
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 42 | 41
participants
  Non serious Infections requiring IV treatment | 4 | 1
  Potential Opportunistic Infections | 5 | 4
  Injection Related Reactions | 2 | 5
  Anaphylaxis | 0 | 0

29. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations Collected by Columbia-Suicide Severity Rating Scale in the DB Period
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool to evaluate suicidal ideation and behavior. Categories have binary responses (yes/no) and include: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation or behavior is indicated by a "yes" answer to any of the listed categories. A score of 0 is assigned if no suicide risk is present. A score of 1 or higher indicates suicidal ideation or behavior.
Time Frame: Baseline and Post-Baseline (up to Week 224)
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo + Baseline Treatment | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 41 | 41
participants
  Baseline: number analyzed (Participants) | 41 | 40
  Baseline | 5 | 12
  Post-Baseline | 2 | 3

30. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies to Satralizumab in the DB Period
Description: Reported here is the percentage of participants with at least one positive anti-drug antibody measurement during the DB period.
Time Frame: Up to approximately Week 224
Population: Participants from SAF who received satralizumab were evaluated for this outcome measure. The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo. Data was summarized together for this outcome measure.
Measure: Number; unit: percentage
Arm/Group | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 41
percentage | 41.5

31. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies to Satralizumab Overall S237 Period
Description: Reported here is the percentage of participants with at least one positive anti-drug antibody measurement during Overall S237 period.
Time Frame: Up to approximately Week 368
Population: as for outcome 30
Measure: Number; unit: percentage
Arm/Group | Satralizumab + Baseline Treatment
Number analyzed (Participants) | 75
percentage
  Treatment-Boosted ADA Patients | 2.7
  Treatment-Induced ADA Patients | 44.0

ADVERSE EVENTS:
Time Frame: Up to 7 years, 9 months, 26 days
Description: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Groups:
- Placebo + Baseline Treatment Double Blind Period: Participants randomized to this arm for the double-blind period received placebo in addition to baseline treatment. The double-blind period ends when either the participant has a treated relapse or the total number of protocol-defined relapses confirmed by the Clinical Endpoint Committee (CEC) reaches 26.
- Satralizumab + Baseline Treatment Double Blind Period: Participants randomized to this arm for the double-blind period received satralizumab in addition to baseline treatment. The double-blind period ends when either the participant has a treated relapse or the total number of protocol-defined relapses confirmed by the Clinical Endpoint Committee (CEC) reaches 26.
- Placebo + Baseline Treatment Open Label Period; Satralizumab + Baseline Treatment Open Label Period: In the open-label extension period, the participant received (with or without baseline treatment) an SC injection of satralizumab at Weeks 0, 2, and 4, and Q4W thereafter, with the last study drug administration on or before 31 December 2021.
- Satralizumab Open-Label Period: In the open-label extension period, the participant received an SC injection of satralizumab at Weeks 0,2, and 4, and Q4W thereafter, in addition to baseline treatment
Arm/Group | Placebo + Baseline Treatment Double Blind Period | Satralizumab + Baseline Treatment Double Blind Period | Placebo + Baseline Treatment Open Label Period | Satralizumab + Baseline Treatment Open Label Period | Satralizumab Open-Label Period
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/32 | 0/39 | 0/1
Serious Adverse Events (participants affected / at risk) | 9/42 | 9/42 | 5/32 | 8/39 | 1/1
Other Adverse Events (participants affected / at risk) | 37/42 | 35/42 | 30/32 | 30/39 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Baseline Treatment Double Blind Period (N=42) | Satralizumab + Baseline Treatment Double Blind Period (N=42) | Placebo + Baseline Treatment Open Label Period (N=32) | Satralizumab + Baseline Treatment Open Label Period (N=39) | Satralizumab Open-Label Period (N=1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuromyelitis optica pseudo relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Baseline Treatment Double Blind Period (N=42) | Satralizumab + Baseline Treatment Double Blind Period (N=42) | Placebo + Baseline Treatment Open Label Period (N=32) | Satralizumab + Baseline Treatment Open Label Period (N=39) | Satralizumab Open-Label Period (N=1)
Anaemia (Blood and lymphatic system disorders) | 5 (8) | 3 (3) | 2 (2) | 5 (7) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 4 (4) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (12) | 6 (10) | 5 (6) | 4 (10) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 (9) | 3 (7) | 1 (1) | 4 (14) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (3) | 1 (1) | 2 (5) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 2 (4) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (8) | 2 (2) | 2 (4) | 2 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (3) | 5 (5) | 3 (5) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 4 (6) | 4 (5) | 3 (3) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (13) | 10 (22) | 11 (49) | 7 (15) | 0 (0)
Oral herpes (Infections and infestations) | 3 (19) | 2 (6) | 4 (42) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (10) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (4) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (12) | 10 (26) | 8 (10) | 8 (36) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 6 (8) | 6 (16) | 5 (23) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (10) | 2 (2) | 2 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (5) | 3 (3) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 10 (28) | 5 (8) | 6 (10) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 3 (3) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 1 (2) | 2 (7) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (6) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (2) | 5 (5) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 2 (6) | 1 (2) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 2 (5) | 1 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocomplementaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (5) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (2) | 2 (8) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte percentage increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Neutrophil percentage increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02028884/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT02028884/SAP_001.pdf